CLINICAL TRIAL: NCT06584461
Title: Lidocaine in Children with Upper Airway Infection Undergoing General Anesthesia: Interventional Controlled Randomized Double Blind Study
Brief Title: Interest of Lidocaine in Children with Upper Airway Infection Undergoing General Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tunis University (Other)
Responsible Party: Principal Investigator, Mehdi Trifa, Full Professor of Anesthesiology and Intensive Care, head chief of the department of Anesthesia and Intensive Care, Tunis University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 092023
Record Dates: First submitted 2024-09-02; First posted 2024-09-04 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Upper Respiratory Tract Infections; Perioperative Respiratory Complications
Keywords: upper respiratory tract infections; IV lidocaine; General anesthesia; children; laryngospasm; bronchospasm; cough; perioperative respiratory complications
MeSH Terms: conditions — Respiratory Tract Infections; Laryngismus; Bronchial Spasm; Cough | interventions — Lidocaine; Pharmaceutical Preparations; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group L: IV Lidocaine Group (Experimental): Participants in this group will receive a volume of weight*0.15 ml intravenous (IV) lidocaine at a dose of 1.5 mg/kg diluted to 10 mg/mL, administered at the induction of anesthesia..
  Interventions: Drug: Lidocaine (drug)
- Group P: Placebo Group (Placebo Comparator): Participants in this group will receive an intravenous placebo (normal saline solution), equivalent in volume (weight*0.15 ml) to the lidocaine group, administered at the induction of anesthesia.
  Interventions: Drug: Saline (NaCl 0,9 %) (placebo)

INTERVENTIONS:
Drug: Lidocaine (drug) — IV lidocaine, administered once during the induction of anesthesia.
  Arms: Group L: IV Lidocaine Group
Drug: Saline (NaCl 0,9 %) (placebo) — IV placebo (normal saline), administered once during the induction of anesthesia.
  Arms: Group P: Placebo Group

SUMMARY:
The goal of this clinical trial is to determine whether intravenous (IV) lidocaine reduces the incidence of perioperative respiratory complications (PRCs) in children with upper respiratory tract infections undergoing general anesthesia. The study will also evaluate the safety of IV lidocaine in this population. The main questions it aims to answer are:

1. Does IV lidocaine lower the incidence of perioperative respiratory complications (e.g., laryngospasm, cough, desaturation) compared to a placebo?
2. What are the side effects associated with the administration of IV lidocaine in these children? Researchers will compare IV lidocaine to a placebo to assess its effectiveness in reducing PRCs.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1 to 14 years.
* American Society of Anesthesiologists (ASA) Physical Status Classification I, II, or III.
* Scheduled or urgent surgery or radiological exploration under general anesthesia.
* Upper respiratory tract infection (URTI) symptoms present for less than 15 days.

Exclusion Criteria:

* Refusal of participation by parents.
* Children on long-term corticosteroid or bronchodilator therapy.
* Contraindications to the use of lidocaine or other drugs used in the protocol.
* Patients who did not adhere to the study protocol.

Ages: 12 Months to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 102 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Incidence of Perioperative Respiratory Complications | Within the first 2 hours post-operation.
  Measure the occurrence of perioperative respiratory complications (e.g., laryngospasm, cough, desaturation, bronchospasm) from the induction of anesthesia until discharge from the recovery room.

SECONDARY OUTCOMES:
Incidence of Side Effects Related to IV Lidocaine | Within the first 24 hours post-operation.
  Measure the occurrence of side effects such as nausea, vomiting, cardiac or neurological toxicity, and signs of anaphylaxis following the administration of IV lidocaine.

CONTACTS AND LOCATIONS:
Locations (1):
- Bechir Hamza Children's Hospital, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: No